CLINICAL TRIAL: NCT05542407
Title: Phase 1 Clinical Trial of ONC201 and Atezolizumab in Obesity-Driven Endometrial Cancer
Brief Title: ONC201 and Atezolizumab in Obesity-Driven Endometrial Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Oncoceutics, Inc. (Industry); National Cancer Institute (NCI) (NIH); Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2036; 5R21CA267584 (NIH)
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer; Metastasis; Endometrioid Endometrial Cancer; Carcinosarcoma; Serous Adenocarcinoma of Endometrium (Diagnosis); Clear Cell Endometrial Carcinoma; Endometrial Endometrioid Adenocarcinoma; Endometrial Mixed Cell Adenocarcinoma
Keywords: Atezolizumab; ONC201; obesity
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasm Metastasis; Carcinosarcoma; Disease; Obesity | interventions — atezolizumab; TIC10 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obese (Experimental): Subjects with BMI > 30 kg/m2
  Interventions: Drug: Atezolizumab; Drug: ONC201
- Non-Obese (Experimental): Subjects with BMI ≤ 29.9 kg/m2
  Interventions: Drug: Atezolizumab; Drug: ONC201

INTERVENTIONS:
Drug: Atezolizumab — 10 mg/kg- 20 mg/kg Atezolizumab will be administered by intravenous, on day 1 of each 21-day cycle.
Drug: ONC201 — 375 mg once weekly - 625 mg ONC201 will be administered orally, once or twice weekly.

SUMMARY:
Endometrial cancer (EC) is the fourth most common cancer in United States women, and alarmingly, the frequency and mortality from EC continues to rise, in part due to the obesity epidemic. Obese women with EC have a 6.3-fold increased risk of death from this disease, as compared to their non-obese counterparts. Patients with advanced/recurrent EC are unlikely to be cured by surgery, conventional chemotherapy (paclitaxel + carboplatin is the standard first-line treatment), radiation, or a combination of these. Thus, new treatments for EC are desperately needed as well as a better understanding of the impact of obesity on EC biology and treatment.

The purpose of this study is to test the safety of a combination of treatments, atezolizumab and ONC201, given based on body weight, to treat endometrial cancer. Using the combination of atezolizumab and ONC201, has not been approved by the Food and Drug Administration (FDA) for the treatment of endometrial cancer. This clinical trial will examine the treatment of atezolizumab + ONC201 in obese and non-obese subjects with metastatic/recurrent EC.

ELIGIBILITY:
In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

Inclusion Criteria

1. Ability to understand and willingness to sign a written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
2. Age ≥ 18 years at the time of consent.
3. ECOG Performance Status of 0, 1, or 2
4. Histologically confirmed metastatic or recurrent EC (endometrioid, carcinosarcoma, serous, clear cell, adeno-squamous and mixed histologies).
5. Subjects must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria
6. Must have radiographic disease progression after at least 1 line of systemic cytotoxic therapy for metastatic disease or with progression within 12 months of completing adjuvant chemotherapy.
7. Life expectancy of at least 3 months.
8. Demonstrate adequate organ function as defined in the table below; all screening labs to be obtained within 72 hours prior to initiating study treatment.

Exclusion Criteria

1. Prior treatment with ONC201.
2. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including antiCTLA-4, and anti PD-L1 therapeutic antibodies
3. Treatment with another investigational agent or participation in another clinical trial within the last 28 days prior to initiating protocol therapy.
4. Subjects who have had chemotherapy or radiotherapy within 4 weeks prior to study treatment or those who have not recovered from adverse events due to agents administered more than 4 weeks prior to initiating protocol therapy.
5. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of protocol therapy Subjects receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
6. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of protocol therapy.
7. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti TNF-agents) within 2 weeks prior to initiation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 58 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2028-02-21 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) | Up to 3 weeks
  The RP2D will be determined based on the incidence of dose-limiting toxicities (DLT)s. A DLT is defined as all grade 3 or above toxicities that are related to study treatment and occur within the first cycle of therapy. Adverse events are assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE). A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate Instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years
  ORR is defined as the proportion of subjects achieving response complete response (CR) or partial response(PR) assessed by RECIST v1.1.
  Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions.
Progression Free Survival (PFS) | Up to 2 years
  PFS is defined as time from first day of treatment until disease progression as defined by RECIST v1.1 or death from any cause.
Overall Survival (OS) | Up to 2 years
  OS is defined as the time of the start of study treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Bae-Jump, MD, PhD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials